CLINICAL TRIAL: NCT03354923
Title: Parent-Child Reciprocity and the Effectiveness of a Parent-Assisted Social Skills Training Program for Adolescents With Autism Spectrum Disorder
Brief Title: Parent-Child Reciprocity and the Effectiveness of PEERS
Acronym: ISR-PEERS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Ofer Golan, Prof. Ofer Golan, Bar-Ilan University, Israel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIU121216
Record Dates: First submitted 2017-01-29; First posted 2017-11-28 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Social Skills; Parent-Child Relational Problem
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate intervention group (Experimental): Immediate PEERS intervention
  Interventions: Behavioral: PEERS intervention
- delayed intervention (Other): delayed PEERS intervention to begin after experimental group
  Interventions: Behavioral: PEERS intervention

INTERVENTIONS:
Behavioral: PEERS intervention — PEERS is a 14-week manualized social skills treatment program that targets the friendship skills of adolescents with ASD. In the Israeli adaptation of PEERS, two meeting were extended. An adolescents group will be held concurrently with the parents group in different rooms. Both groups will begin the session with homework review, followed by a didactic social skills lesson, utilizing the teaching methods of modeling and role-playing. In order to practice the newly learned social skills,a behavioral rehearsal interaction will be assigned in the adolescents group. Finally,Socialization homework assignments designed to address further mastery and generalization of newly learned skills within the natural social environment will be assigned too.

SUMMARY:
Early adolescence marks a significant development in teens' social abilities, shifting from play to conversation-based activities, and having stronger and more intimate friendships. Parents contribute to this shift by practicing reciprocal social interaction with their teens.

For teens with Autism Spectrum Disorder (ASD) this shift in their peers' social abilities extends their characteristic social deficits even further. Social skills deficits in individuals with ASD are associated with poor adaptive functioning and increased psychopathology. Parents play a pivotal role in caring for and tutoring their children with ASD into adulthood. However, the effect parent-teen reciprocity has on the social skills of adolescents with ASD has not been tested. Furthermore, whereas parent-child reciprocity predicted intervention outcome in young children with ASD, no study has examined this effect in teens with ASD.

The proposed study aims to test these questions using the Program for the Education and Enrichment of Relational Skills (PEERS), an evidence-based parent-assisted social skills training program for teens with ASD.

DETAILED DESCRIPTION:
Entering adolescence is a significant milestone in the development of socialization. Same-sex friendships and "best friends", developed during childhood, become more intensive, reciprocal, and intimate. In addition, social networks evolve and become more central for adolescents. Social interaction moves in adolescence from focusing on game playing to conversation focused interaction. Teens begin to exhibit dialogical skills, including the capacity to acknowledge others' opinions and emotions; view oneself in someone else's position; discuss disagreements with empathy while maintaining positive affect; and engage in a give-and-take, fluent, and non-constricted exchange while maintaining an autonomous stance. The consolidation of close friendships requires for teens to learn to dialogue joint positive plans as well as interpersonal conflicts within the relationship. Parents, through their relationships with their teens, can provide them with opportunities to learn, experience, and practice the dialogical skills needed for social functioning. Parental contribution to teens' dialogical skills is possible despite the differences between parent-teen and teen-peers interactions, since interaction in both kinds of relationships requires reciprocity .

Reciprocity is defined as the capacity to engage in social exchange that integrates inputs from multiple partners into a unified social event. It involves an ongoing process of awareness to- and interpretation of- the emotional and interpersonal cues of others, followed by an appropriate response that enables a smooth continuation of the social interaction. Parent-child reciprocity is a key element of early social relationships, which sets the foundation for social collaboration, empathy, and pro-social behavior. Developmental studies have demonstrated how early parent-child reciprocity predicts social adaptive functioning in adolescence, whereas intrusive, controlling parenting is associated with poorer social outcomes, such as affiliations with deviant friends. Adolescents gain from productive reciprocity with the parent, as it gives them an opportunity to express their individuation vis-a-vis the parental stance, and to practice important perspective taking, exchanging information, negotiation, and conflict resolution skills in a secure, enabling environment. The proposed study aims to examine the effect parent-teen reciprocity has on adolescents with an Autism Spectrum Disorder. Autism Spectrum Disorder (ASD) is a neuro-developmental condition, characterized by social communication deficits and restricted and repetitive behavior patterns. ASD symptoms vary in severity (e.g. from total lack of social initiative and extreme difficulty tolerating change, to an awkward social approach and difficulties adapting behavior do the social context), which may be related to different levels of functioning. In addition, ASD can involve intellectual impairment and comorbid psychopathology, that may further hamper independent functioning . Despite positive effects of early intervention social deficits in ASD persist throughout the lifespan even for higher functioning individuals .

For many individuals with ASD, adolescence is a particularly troubling period, characterized by enhanced motivation for social relationships, but at the same time, by increased realization of the difficulties they encounter when interacting with peers and their lack of knowledge and experience in friend-making . As they attempt to integrate socially, adolescents with ASD experience more negative social outcomes (e.g., fewer friends, little support from classmates, limited involvement in social activities, and increased peer rejection) compared to adolescents with other developmental disabilities or typically developing teens. Due to their social-communication deficits as well as their social naivety, adolescents with ASD are also more exposed to bullying, reflected in high rates of victimization and perpetration.

Parents play a pivotal role in caring for their child with ASD. Due to the developmental delays and social isolation of individuals with ASD, parents continue to care for their children into adolescence and adulthood, often as the only carers . Because of their central supportive role in their children's lives, research has attempted to highlight parental factors that may predict the quality of parent-child relationships as well as child outcomes. Most studies observing such parental factors have focused on parents of toddlers and preschoolers, associating parental resolution of the child's diagnosis, parental insightfulness into the experience of the child, and parental sensitivity, with child's secure attachment. Studies of parents' relationship with their older offspring linked maternal pessimism to poorer relationships with sons/daughters with ASD , and maternal warmth and praise with lower levels of internalizing and externalizing symptoms in adolescents and adults with ASD. However, these studies are based on self and parental report rather than on behavioral observation, and did not examine parent-teen reciprocity.

Examinations of the effects of parent-child reciprocity on children with ASD have mostly focused on young children. Our own work showed parent-child reciprocity is associated with improved emotion regulation and lower negative emotionality as well as with increased levels of oxytocin in children with ASD. On the other hand, controlling, intrusive parenting was associated with externalizing behavior problems in children and adolescents with ASD. Parent-child reciprocity has also been shown to predict higher social skills of children with ASD and to mediate the relation between child's level of functioning and social skills. The contribution of parent-child reciprocity to the child's intervention related progress has been addressed in some intervention studies for toddlers and pre-schoolers with ASD , revealing parent-child reciprocity mediates the effect of social communication interventions in this young age group. However, an examination of parentadolescent reciprocity in ASD, as a predictor of teen outcome is still needed.

The complexity of the parental role in adolescence is greater and more stressful when parenting teens with ASD . The need for greater parental input into the nature of social interaction, the new themes of intimacy and sexuality brought upon by puberty, and the parental wish to protect their teens from exclusion and bullying may bring parents to be more controlling, and even intrusive in their interaction with their teens . However, as described above, parent-teen reciprocity is important in developing teens' appropriate social reciprocity with peers. Hence, the ability of parents to be more reciprocal and less intrusive in their interaction with their teens is expected to predict teens' social skills and reciprocity with peers. Furthermore, parent-teen reciprocity is expected to play a part in the ability of teens and parents to gain from interventions targeting social skills, such as parent-assisted social skills groups.

PEERS Intervention: Social skills groups are common interventions for people with ASD, especially those with average to above-average cognitive skills . However, the majority of social skills training programs have focused on children aged 7-12, and few studies have examined the benefit of such groups for adolescents with ASD . Furthermore, few Randomized Controlled Trials (RCTs) have examined the effectiveness of social skills training for those with ASD. The proposed study aims to conduct the first RCT of a social skills training program for adolescents with ASD in Israel, using the well-established Program for the Education and Enrichment of Relational Skills (PEERS). PEERS , is a parent-assisted, manualized social skills training program for high-functioning adolescents with ASD, addressing crucial areas of social functioning for adolescents (see methods for a description). Ecologically valid skills for making and maintaining friends are taught using psychoeducational and cognitive-behavioral treatment techniques. Parents learn how to be social coaches to their teens in a separate group, running in parallel to the teens' group. Teens practice the taught skills in between sessions. Parents, as social coaches, are expected to supervise their teens' treatment fidelity, and in addition to practice the taught skills with their teens (e.g., running a two-way conversation, noticing the others' non-verbal cues, etc.). In North America, PEERS has been evaluated using RCTs, with its efficacy established for improving a variety of social skills in adolescents, including social skills knowledge, social responsiveness, social communication, social cognition, social awareness, social motivation, assertion, cooperation, and responsibility . PEERS related gains were maintained even 5 years post intervention. PEERS treatment effects have also been reflected in changes in the social brain as revealed through biomarkers of treatment outcome using EEG . A first cross-cultural validation study of PEERS in South Korea, yielded a significant improvement in teens' social skills knowledge, interpersonal skills, play/leisure skills, and a decrease in teens' autism symptoms and depression, as well as parents' anxiety. Recently, two preintervention child factors; parental report on teens' social skills, and teens' self-awareness of their popularity, were found to predict PEERS intervention outcome. PEERS positive effects on parents' self-efficacy have also been reported. However, although PEERS relies on parents as social coaches, the effect of parent-teen reciprocity on PEERS outcome has not been examined. As in everyday life, parents have a complex role in PEERS: On one hand, supervising their teens' work may call for more controlling, intrusive parenting. On the other hand, in order to effectively practice the taught social skills with their teens (and to meet the program's goals), parents and teens need to reciprocally collaborate. The use of reciprocity and intrusiveness in parent-teen interaction could therefore mediate the effect of PEERS on teens' social skills. In addition, since PEERS also teaches parents how to be less intrusive and more reciprocal with their teens, an improvement in parent-teen reciprocity is expected

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide informed assent
* Diagnosed with ASD (high functioning)
* IQ > 80

Exclusion Criteria:

* Intellectual Disability
* History of significant head injury or neurological illness
* Current diagnosis of substance dependence

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Parent-Adolescent reciprocity paradigm at 4 and 8 months | Day 0, 4 months and 8 months
  This paradigm is designed to test dyadic reciprocity between a parent and an adolescent. Adolescents will be observed in three 10-minute discussions (one positive, one support giving and one negative) with the parent who serves as their PEERS coach: In the positive discussion, parent and teen will be asked to plan a fun outing together. In the support giving the parent and child take turns and each tells the other something sad/disappointing that happened to him/her outside the relationship (with friends, boss, etc.) and the other gives support. After five minutes partners change roles. In the negative discussion they will be asked about a common conflict between them and negotiate it. The three discussions will be videotaped and coded using the Coding Interactive Behavior manual (Feldman, 1998). The CIB is a global rating system for social interactions that includes 52 codes rated on a scale of 1 to 5 which are aggregated into several composites
Change from baseline Contextual Assessment of Social Skills at 4 and 8 months | Day 0, 4 months and 8 months
  The CASS is a live role-play assessment of conversational skills developed for adolescents with high-functioning ASD. Conversational skills are assessed via behavioral coding of two semi-structured role-plays (with an interested companion and with a bored companion) and scores on a conversation rating scale. Behaviors coded during the role plays include asking questions, topic changes, vocal expressiveness, gestures, positive affect, posture, kinesics arousal, social anxiety, involvement in the conversation, quality of rapport, and an overall score. Psychometric properties of the CASS are good, with mean internal consistency of .83 and mean inter-rater reliability of .68. The CASS was reported as a sensitive measure of change in an evaluation of a social skills program for young adults with ASD (White, Scarpa, Conner, Maddox, & Bonete, 2014).

SECONDARY OUTCOMES:
Change from baseline Social Responsiveness Scale at 4 and 8 months | Day 0, 4 months and 8 months
  The SRS is a 65-item rating scale measuring the severity of autism spectrum symptoms as they occur in natural social settings. Completed by parents and teachers, it is appropriate for use with children from 4 to 18 years of age. Scales include social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits. The SRS has been shown to be sensitive to changes in social functioning among children with ASD (Wood et al., 2009). Internal consistency for SRS scales varies between 0.91-0.97, test-retest reliability 0.84-0.97 and interrater reliability 0.74-0.95 (Bolte, Poustka, & Constantino, 2008).
Change from baseline The Social Skills Improvement System at 4 and 8 months | Day 0, 4 months and 8 months
  The SSIS is a standardized rating scale that assesses global social competence for children 3 to 18 years. Designed to assess social skills change after treatment, it utilizes a multi-informant approach, allowing parents, teachers, and students to evaluate target social behaviors including communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. Targeted problem behaviors include externalizing behaviors and bullying. Internal consistency for the SSIS ranges from .92 to .97, test-retest reliability from .77 to .87, inter-rater reliability from .50 to .68.
Change from baseline Friendship Qualities Scale | Day 0, 4 months and 8 months
  The FQS is an adolescent self-report measure of the quality of best friendships. It is composed of 23-items on a scale of 0-4. The items fall into five categories: Closeness, Companionship, Conflict, Helpfulness, and Security. The FQS has good internal consistency, with alpha coefficients ranging between .71 and .86 across all five categories.
Change from baseline Quality of Play Questionnaire at 4 and 8 months | Day 0, 4 months and 8 months
  The QPQ is a measure completed by adolescents (QPQ-A) and parents (QPQ-P) in which the quality of the adolescent's last get-together and the frequency of weekly get-togethers with peers are assessed. The scales on the QPQ have been shown to discriminate individuals referred to social skills training from a general community sample using a cut point of > 3.5 on the Conflict Scale and a cut point of < 2.5 on the frequencies of get-togethers.
Change from baseline Test of Adolescent Social Skills Knowledge at 4 and 8 months | Day 0, 4 months and 8 months
  The TAASK is a criterion referenced measure designed to assess adolescent knowledge of the specific social skills taught during the PEERS treatment. Two items are derived from each of the PEERS didactic lessons making a total of 26 forced-choice items.
Change from baseline Vineland Adaptive Behaviors Scales II at 4 and 8 months | Day 0, 4 months and 8 months
  The VABS II is a parent interview regarding a child communication, social, motor and daily living skills based on the report of primary caregivers from which a standardized composite score of adaptive function is calculated.
Change from baseline Loneliness and Social Dissatisfaction Questionnaire at 4 and 8 months | Day 0, 4 months and 8 months
  The LSDQ is a 24-item, standardized self-report measure that assesses global feelings of loneliness and social adequacy and inadequacy. It has been validated with typically developing youth, as well as youth with intellectual disabilities and learning disabilities.
Change from baseline Beck Depression Inventory II at 4 and 8 months | Day 0, 4 months and 8 months
  The BDI-II is a 21 items self-administered questionnaire consisting of 21 items that assess the severity of symptoms and attitudes related to depression. The questionnaire identifies the presence and severity of symptoms consistent with the criteria of the DSM-V. The sum of the scores obtained in each item results in a total score when 14-19 is considered as mild, 20-28 moderate and 29-63 is considered as severe symptoms of depression.
Change from baseline Autism Spectrum Quotient at 4 and 8 months | Day 0, 4 months and 8 months
  The AQ is 50 item, self-reported questionnaire measuring the degree to which an adult with normal intelligence has the traits associated with the autistic spectrum. The cut of score which indicates the person has clinically significant levels of autistic traits is 32 or more. The AQ is a well-known screening instrument for autism spectrum disorder
Change from baseline Empathy Quotient at 4 and 8 months | Day 0, 4 months and 8 months
  The EQ is a 60 item, valid self-assessment questionnaire measuring empathy levels in adults with normal intelligence. The scales of EQ are 0-80 with the cut off score of 30. The EQ is used as a screening instrument for autism spectrum disorder.
Change from baseline Parenting Stress Index Short Form at 4 and 8 months | Day 0, 4 months and 8 months
  . The PSI/SF is a 36 item, self-reported questionnaire for parents measuring the levels of stress in the parent-child relationship and identifies the presence of dysfunctional parenting. This instrument has 4 subscales: Defensive responsive, Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child. Child and Parent domains combine to form the Total Stress Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Irit Mor, MD, Principal Investigator — Association for Children at Risk
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hartup WW. Adolescents and their friends. New Dir Child Dev. 1993 Summer;(60):3-22. doi: 10.1002/cd.23219936003. No abstract available. PMID 8414122
- [Background] Lempers JD, Clark-Lempers DS. Young, middle, and late adolescents' comparisons of the functional importance of five significant relationships. J Youth Adolesc. 1992 Feb;21(1):53-96. doi: 10.1007/BF01536983. PMID 24263682
- [Background] Paul R. Promoting social communication in high functioning individuals with autistic spectrum disorders. Child Adolesc Psychiatr Clin N Am. 2003 Jan;12(1):87-106, vi-vii. doi: 10.1016/s1056-4993(02)00047-0. PMID 12512400
- [Background] Constantino JN, Davis SA, Todd RD, Schindler MK, Gross MM, Brophy SL, Metzger LM, Shoushtari CS, Splinter R, Reich W. Validation of a brief quantitative measure of autistic traits: comparison of the social responsiveness scale with the autism diagnostic interview-revised. J Autism Dev Disord. 2003 Aug;33(4):427-33. doi: 10.1023/a:1025014929212. PMID 12959421
- [Background] Feldman R. Mother-infant synchrony and the development of moral orientation in childhood and adolescence: direct and indirect mechanisms of developmental continuity. Am J Orthopsychiatry. 2007 Oct;77(4):582-97. doi: 10.1037/0002-9432.77.4.582. PMID 18194038
- [Background] Feldman R, Bamberger E, Kanat-Maymon Y. Parent-specific reciprocity from infancy to adolescence shapes children's social competence and dialogical skills. Attach Hum Dev. 2013;15(4):407-23. doi: 10.1080/14616734.2013.782650. Epub 2013 Apr 2. PMID 23544455
- [Background] Soenens, B., Vansteenkiste, M., Smits, I., Lowet, K., & Goossens, L. (2007). The role of intrusive parenting in the relationship between peer management strategies and peer affiliation. Journal of Applied Developmental Psychology, 28(3), 239-249.
- [Background] McElhaney, K. B., Allen, J. P., Stephenson, J. C., & Hare, A. L. (2009). Attachment and Autonomy during Adolescence. In Handbook of Adolescent Psychology. Hoboken, NJ, USA: John Wiley & Sons, Inc.
- [Background] Russell, A., Pettit, G. S., & Mize, J. (1998). Horizontal Qualities in Parent-Child Relationships: Parallels with and Possible Consequences for Children's Peer Relationships. Developmental Review, 18(3), 313-352
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders. American Psychiatric Association.
- [Background] Dawson G, Zanolli K. Early intervention and brain plasticity in autism. Novartis Found Symp. 2003;251:266-74; discussion 274-80, 281-97. PMID 14521198
- [Background] Howlin, P. (2004). Autism and Asperger syndrome: Preparing for adulthood. London: Routledge.
- [Background] Tantam D. The challenge of adolescents and adults with Asperger syndrome. Child Adolesc Psychiatr Clin N Am. 2003 Jan;12(1):143-63, vii-viii. doi: 10.1016/s1056-4993(02)00053-6. PMID 12512403
- [Background] Haddad J. Social skills for teenagers with developmental and autism spectrum disorders: The PEERS treatment manual. J Child Adolesc Ment Health. 2013;25(1):93-4. doi: 10.2989/17280583.2013.802447. No abstract available. PMID 25860311
- [Background] Renno P, Wood JJ. Discriminant and convergent validity of the anxiety construct in children with autism spectrum disorders. J Autism Dev Disord. 2013 Sep;43(9):2135-46. doi: 10.1007/s10803-013-1767-1. PMID 23354538
- [Background] Sofronoff K, Dark E, Stone V. Social vulnerability and bullying in children with Asperger syndrome. Autism. 2011 May;15(3):355-72. doi: 10.1177/1362361310365070. Epub 2011 Mar 23. PMID 21430018
- [Background] Gerhardt, P. F., & Lainer, I. (2011). Addressing the Needs of Adolescents and Adults with Autism: A Crisis on the Horizon. Journal of Contemporary Psychotherapy, 41(1), 37-45.
- [Background] Milshtein S, Yirmiya N, Oppenheim D, Koren-Karie N, Levi S. Resolution of the diagnosis among parents of children with autism spectrum disorder: associations with child and parent characteristics. J Autism Dev Disord. 2010 Jan;40(1):89-99. doi: 10.1007/s10803-009-0837-x. Epub 2009 Jul 31. PMID 19644747
- [Background] Oppenheim D, Koren-Karie N, Dolev S, Yirmiya N. Maternal insightfulness and resolution of the diagnosis are associated with secure attachment in preschoolers with autism spectrum disorders. Child Dev. 2009 Mar-Apr;80(2):519-27. doi: 10.1111/j.1467-8624.2009.01276.x. PMID 19467008
- [Background] Orsmond GI, Seltzer MM, Greenberg JS, Krauss MW. Mother-child relationship quality among adolescents and adults with autism. Am J Ment Retard. 2006 Mar;111(2):121-37. doi: 10.1352/0895-8017(2006)111[121:MRQAAA]2.0.CO;2. PMID 16466284
- [Background] Smith LE, Greenberg JS, Seltzer MM, Hong J. Symptoms and behavior problems of adolescents and adults with autism: effects of mother-child relationship quality, warmth, and praise. Am J Ment Retard. 2008 Sep;113(5):387-402. doi: 10.1352/2008.113:387-402. PMID 18702558
- [Background] Hirschler-Guttenberg Y, Golan O, Ostfeld-Etzion S, Feldman R. Mothering, fathering, and the regulation of negative and positive emotions in high-functioning preschoolers with autism spectrum disorder. J Child Psychol Psychiatry. 2015 May;56(5):530-9. doi: 10.1111/jcpp.12311. Epub 2014 Aug 14. PMID 25123380
- [Background] Feldman R, Golan O, Hirschler-Guttenberg Y, Ostfeld-Etzion S, Zagoory-Sharon O. Parent-child interaction and oxytocin production in pre-schoolers with autism spectrum disorder. Br J Psychiatry. 2014 Aug;205(2):107-12. doi: 10.1192/bjp.bp.113.137513. Epub 2014 May 22. PMID 24855128
- [Background] Maljaars J, Boonen H, Lambrechts G, Van Leeuwen K, Noens I. Maternal parenting behavior and child behavior problems in families of children and adolescents with autism spectrum disorder. J Autism Dev Disord. 2014 Mar;44(3):501-12. doi: 10.1007/s10803-013-1894-8. PMID 23881094
- [Background] Haven EL, Manangan CN, Sparrow JK, Wilson BJ. The relation of parent-child interaction qualities to social skills in children with and without autism spectrum disorders. Autism. 2014 Apr;18(3):292-300. doi: 10.1177/1362361312470036. Epub 2013 Sep 26. PMID 24072662
- [Background] Kasari C, Gulsrud AC, Wong C, Kwon S, Locke J. Randomized controlled caregiver mediated joint engagement intervention for toddlers with autism. J Autism Dev Disord. 2010 Sep;40(9):1045-56. doi: 10.1007/s10803-010-0955-5. PMID 20145986
- [Background] Rogers SJ, Estes A, Lord C, Vismara L, Winter J, Fitzpatrick A, Guo M, Dawson G. Effects of a brief Early Start Denver model (ESDM)-based parent intervention on toddlers at risk for autism spectrum disorders: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Oct;51(10):1052-65. doi: 10.1016/j.jaac.2012.08.003. Epub 2012 Aug 28. PMID 23021480
- [Background] Fong, L., Wilgosh, L., & Sobsey, D. (1993). The Experience of Parenting an Adolescent with Autism. International Journal of Disability, Development and Education, 40(2), 105-113.
- [Background] Reaven J, Blakeley-Smith A, Culhane-Shelburne K, Hepburn S. Group cognitive behavior therapy for children with high-functioning autism spectrum disorders and anxiety: a randomized trial. J Child Psychol Psychiatry. 2012 Apr;53(4):410-9. doi: 10.1111/j.1469-7610.2011.02486.x. PMID 22435114
- [Background] Reichow B, Steiner AM, Volkmar F. Social skills groups for people aged 6 to 21 with autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008511. doi: 10.1002/14651858.CD008511.pub2. PMID 22786515
- [Background] Cappadocia, M. C., & Weiss, J. A. (2011). Review of social skills training groups for youth with Asperger Syndrome and High Functioning Autism. Research in Autism Spectrum Disorders, 5(1), 70-78.
- [Background] Laugeson EA, Frankel F, Gantman A, Dillon AR, Mogil C. Evidence-based social skills training for adolescents with autism spectrum disorders: the UCLA PEERS program. J Autism Dev Disord. 2012 Jun;42(6):1025-36. doi: 10.1007/s10803-011-1339-1. PMID 21858588
- [Background] Schohl KA, Van Hecke AV, Carson AM, Dolan B, Karst J, Stevens S. A replication and extension of the PEERS intervention: examining effects on social skills and social anxiety in adolescents with autism spectrum disorders. J Autism Dev Disord. 2014 Mar;44(3):532-45. doi: 10.1007/s10803-013-1900-1. PMID 23893101
- [Background] Laugeson EA, Frankel F, Mogil C, Dillon AR. Parent-assisted social skills training to improve friendships in teens with autism spectrum disorders. J Autism Dev Disord. 2009 Apr;39(4):596-606. doi: 10.1007/s10803-008-0664-5. Epub 2008 Nov 18. PMID 19015968
- [Background] Mandelberg, J., Laugeson, E. A., Cunningham, T. D., Ellingsen, R., Bates, S., & Frankel, F. (2014). Long-Term Treatment Outcomes for Parent-Assisted Social Skills Training for Adolescents with Autism Spectrum Disorders: The UCLA PEERS Program. Journal of Mental Health Research in Intellectual Disabilities, 7(1), 45-73
- [Background] Van Hecke AV, Stevens S, Carson AM, Karst JS, Dolan B, Schohl K, McKindles RJ, Remmel R, Brockman S. Measuring the plasticity of social approach: a randomized controlled trial of the effects of the PEERS intervention on EEG asymmetry in adolescents with autism spectrum disorders. J Autism Dev Disord. 2015 Feb;45(2):316-35. doi: 10.1007/s10803-013-1883-y. PMID 23812665
- [Background] Yoo HJ, Bahn G, Cho IH, Kim EK, Kim JH, Min JW, Lee WH, Seo JS, Jun SS, Bong G, Cho S, Shin MS, Kim BN, Kim JW, Park S, Laugeson EA. A randomized controlled trial of the Korean version of the PEERS((R)) parent-assisted social skills training program for teens with ASD. Autism Res. 2014 Feb;7(1):145-61. doi: 10.1002/aur.1354. Epub 2014 Jan 9. PMID 24408892
- [Background] Chang YC, Laugeson EA, Gantman A, Ellingsen R, Frankel F, Dillon AR. Predicting treatment success in social skills training for adolescents with autism spectrum disorders: the UCLA Program for the Education and Enrichment of Relational Skills. Autism. 2014 May;18(4):467-70. doi: 10.1177/1362361313478995. Epub 2013 Oct 9. PMID 24108192
- [Result] Pickles A, Harris V, Green J, Aldred C, McConachie H, Slonims V, Le Couteur A, Hudry K, Charman T; PACT Consortium. Treatment mechanism in the MRC preschool autism communication trial: implications for study design and parent-focussed therapy for children. J Child Psychol Psychiatry. 2015 Feb;56(2):162-70. doi: 10.1111/jcpp.12291. Epub 2014 Jul 8. PMID 25039961
- [Result] Feldman, R. (1998). Coding interactive behavior. Unpublished Manual, 1-54.
- [Result] Ratto AB, Turner-Brown L, Rupp BM, Mesibov GB, Penn DL. Development of the Contextual Assessment of Social Skills (CASS): a role play measure of social skill for individuals with high-functioning autism. J Autism Dev Disord. 2011 Sep;41(9):1277-86. doi: 10.1007/s10803-010-1147-z. PMID 21287253
- [Result] Wood JJ, Drahota A, Sze K, Har K, Chiu A, Langer DA. Cognitive behavioral therapy for anxiety in children with autism spectrum disorders: a randomized, controlled trial. J Child Psychol Psychiatry. 2009 Mar;50(3):224-34. doi: 10.1111/j.1469-7610.2008.01948.x. PMID 19309326
- [Result] Gresham, F., & Elliott, S. (2008). Social skills improvement system (SSIS) rating scales. Bloomington, MN: Pearson.
- [Result] Sparrow SS, Cicchetti DV. Diagnostic uses of the Vineland Adaptive Behavior Scales. J Pediatr Psychol. 1985 Jun;10(2):215-25. doi: 10.1093/jpepsy/10.2.215. No abstract available. PMID 4020603
- [Result] Asher, S. R., Hymel, S., & Renshaw, P. D. (1984). Loneliness in Children. Child Development, 55(4), 1456.
- [Result] Beck, A. T., Steer, R. A., & Brown, G. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Result] Baron-Cohen S, Wheelwright S, Skinner R, Martin J, Clubley E. The autism-spectrum quotient (AQ): evidence from Asperger syndrome/high-functioning autism, males and females, scientists and mathematicians. J Autism Dev Disord. 2001 Feb;31(1):5-17. doi: 10.1023/a:1005653411471. PMID 11439754
- [Result] Baron-Cohen S, Wheelwright S. The empathy quotient: an investigation of adults with Asperger syndrome or high functioning autism, and normal sex differences. J Autism Dev Disord. 2004 Apr;34(2):163-75. doi: 10.1023/b:jadd.0000022607.19833.00. PMID 15162935
- [Result] Abidin, R. R. (1990). Parenting stress index-short form. Charlottesville, VA: Pediatric Psychology Press.
- [Result] Frankel F, Mintz J. Maternal Reports of Play Dates of Clinic Referred and Community Children. J Child Fam Stud. 2011 Oct;20(5):623-630. doi: 10.1007/s10826-010-9437-9. Epub 2010 Nov 13. PMID 22003278
- [Result] Laugeson, E. A., & Frankel, F. (unpublished). Test of adolescent social skills knowledge-revised. (Available from UCLA Parenting and Children's Friendship Program, 300 Medical Plaza, Los Angeles, CA 90095, USA).